CLINICAL TRIAL: NCT01628406
Title: Patient Registry of the Neurosurgery Department.
Acronym: patregNCH
Status: Unknown | Type: Observational
Last Known Status: Enrolling by invitation
Sponsor: University of Zurich (Other)
Responsible Party: Sponsor
Other Study IDs: patregNCH
Record Dates: First submitted 2012-06-21; First posted 2012-06-26 (Estimated); Last update posted 2023-12-14 (Actual); Status verified 2023-12

CONDITIONS: Patients Treated at the Neurosurgery Department

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 10 Years

GROUPS / COHORTS (1):
- Patients treated at the neurosurgery department: Patients treated at the neurosurgery department
  Interventions: Procedure: Treatment at the neurosurgery departement

INTERVENTIONS:
Procedure: Treatment at the neurosurgery departement — Treatment at the neurosurgery departement

SUMMARY:
The investigators record all indications, treatments and outcomes from patients treated at the Neurosurgery Department.

* Trial with surgical intervention

ELIGIBILITY:
Inclusion criteria:

All patients treated at the Neurosurgery Department

Exclusion criteria:

None

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: All patients treated at the Neurosurgery Department
Sampling Method: Non-Probability Sample
Enrollment: 18000 (Estimated)
Dates: Start 2012-06; Primary Completion 2025-12 (Estimated); Study Completion 2025-12 (Estimated)

PRIMARY OUTCOMES:
neurological outcome | 1 year
  validated scales like KPSS or NIHSS
social outcome | 1 year
  e.g. activity of daily living, employment status

CONTACTS AND LOCATIONS:
Overall Officials: Johannes Sarnthein, Prof Dr, Principal Investigator — University Hospital Zurich, Division of Neurosurgery; Luca Regli, Prof Dr, Principal Investigator — University Hospital Zurich, Division of Neurosurgery
Locations (1):
- University Hospital Zurich, Neurosurgery, Zurich, Canton of Zurich, Switzerland

REFERENCES:
- [Result] Sarnthein J, Staartjes VE, Regli L; Neurosurgery-Registry consortium. Neurosurgery outcomes and complications in a monocentric 7-year patient registry. Brain Spine. 2022 Jan 19;2:100860. doi: 10.1016/j.bas.2022.100860. eCollection 2022. PMID 36248111
- [Derived] Staartjes VE, Serra C, Regli L. In Reply: Safety and Effectiveness of an Enhanced Recovery Protocol in Patients Undergoing Burr Hole Evacuation for Chronic Subdural Hematoma. Neurosurgery. 2025 Jan 1;96(1):e16-e17. doi: 10.1227/neu.0000000000003235. Epub 2024 Oct 24. No abstract available. PMID 39445855